CLINICAL TRIAL: NCT05770713
Title: Treatment Patterns And Clinical Outcomes Among Patients Receiving CDK4/6 Inhibitors Combinations For HR+/HER2- Advanced/Metastatic Breast Cancer In A Canadian Real World Setting
Brief Title: A Real-life Study to Learn About the Use and Effects of the CDK4/6 Inhibitors in Canadian Patients With Breast Cancer.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481178
Record Dates: First submitted 2023-03-05; First posted 2023-03-15 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: metastatic breast cancer; advanced breast cancer; HR+/HER2-
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Female patients with HR+/HER2- ABC/MBC who received a CDK4/6i based therapy for their ABC/MBC.: Female patients who received an oral treatment of CDK4/6i based therapy for their ABC/MBC.

SUMMARY:
CDK4/6 inhibitors are approved medicines indicated for the treatment of a kind of advanced/metastatic breast cancer, called hormone receptors positive (HR+)/ Human epidermal growth factor receptor 2 negative (HER2-) disease. They are given orally in combination with hormonal therapies.

The purpose of this study is to better understand how the CDK4/6 inhibitors combinations are used in real-life conditions and their clinical impact for the treatment of Canadian patients affected by (HR+)/ (HER2-) advanced breast cancer (ABC) or metastatic breast cancer (MBC).

Female patients aged 18 years old or more presenting the following conditions will be selected for the study:

* HR+/HER2- breast cancer diagnosis with confirmed metastatic or advanced disease
* Diagnosis of ABC/MBC between 01 January 2016 and 01 July 2021
* Treatment with CDK4/6 inhibitor

Information will be collected from one single Canadian institution, on each selected real-life patient treated with CDK4/6 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* HR+/HER2- breast cancer diagnosis with confirmed metastatic or advanced disease
* Diagnosed with ABC/MBC between 01 Jan 2016 and 01 July 2021
* Treatment with CDK4/6 inhibitor

Exclusion Criteria:

* Patient does not have ABC/MBC
* Patient has indicated HR- or HER2+ status
* Patient received a CDK4/6i as part of a clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female patients diagnosed with HR+/HER2- ABC/MBC who received a CDK4/6 inhibitor at Sinai Health, Canada during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Canada, Kirkland, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with hormone receptor-positive (HR+) and human epidermal growth factor receptor 2 negative (HER2)- advanced/metastatic breast cancer (ABC/MBC) between 01-Jan-2016 to 01-Jul-2021 and received a cyclin-dependent kinase 4 and 6 inhibitor (CDK4/6i) at Sinai Health were included in this retrospective study. Data were extracted from electronic health records until 01-Oct-2021. Available data was evaluated from 12-Oct-2022 to 28-Feb-2023 (approximately 4.5 months).
Pre-assignment Details: A total of 48 female participants were included in this study.
Groups:
- HR+/HER2- ABC/MBC Participants: Participants with HR+/HER2- advanced/metastatic breast cancer who received treatment with CDK4/6 inhibitors) at Sinai Health between 01-Jan-2016 to 01-Oct-2021 were observed in this retrospective study.
Period: Overall Study
Arm/Group | HR+/HER2- ABC/MBC Participants
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Arm/Group | HR+/HER2- ABC/MBC Participants
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified According to Treatment Pattern
Description: Number of participants according to the treatment patterns for first line, second line and third line were reported in this outcome measure. CDK4/6i included abemaciclib, palbociclib and ribociclib. Endocrine therapy (ET) included anastrozole, exemestane, fulvestrant, letrozole and tamoxifen. Chemotherapy included capecitabine, cisplatin, cyclophosphamide, docetaxel, doxorubicin, eribulin, gemcitabine and paclitaxel.
Time Frame: From date of ABC/MBC diagnosis until date of death, date of last follow-up or the end of the study period, whichever came first (maximum follow-up of 67.6 months); available data evaluated over approximately 4.5 months of this retrospective study
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study. Here "Number Analyzed" refers to the number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | HR+/HER2- ABC/MBC Participants
Number analyzed (Participants) | 48
Participants
  1st line: Palbociclib + ET | 30
  1st line: Palbociclib + ET + goserelin | NA — Data was not reported for observations including <=5 participants in accordance with hospital data privacy regulations in place at Sinai Health.
  1st line: Other CDK 4/6i + ET | NA — Data was not reported for observations including <=5 participants in accordance with hospital data privacy regulations in place at Sinai Health.
  1st line: Other CDK 4/6i + ET + goserelin | NA — Data was not reported for observations including <=5 participants in accordance with hospital data privacy regulations in place at Sinai Health.
  1st line: ET | NA — Data was not reported for observations including <=5 participants in accordance with hospital data privacy regulations in place at Sinai Health.
  1st line: Chemotherapy | 7
  2nd line: Palbociclib + ET: number analyzed (Participants) | 21
  2nd line: Palbociclib + ET | NA — Data was not reported for observations including <=5 participants in accordance with hospital data privacy regulations in place at Sinai Health.
  2nd line: Palbociclib + ET + goserelin: number analyzed (Participants) | 21
  2nd line: Palbociclib + ET + goserelin | NA — Data was not reported for observations including <=5 participants in accordance with hospital data privacy regulations in place at Sinai Health.
  2nd line: Other CDK 4/6i + ET: number analyzed (Participants) | 21
  2nd line: Other CDK 4/6i + ET | 7
  2nd line: Other CDK 4/6i + ET + goserelin: number analyzed (Participants) | 21
  2nd line: Other CDK 4/6i + ET + goserelin | NA — Data was not reported for observations including <=5 participants in accordance with hospital data privacy regulations in place at Sinai Health.
  2nd line: Alpelisib + ET: number analyzed (Participants) | 21
  2nd line: Alpelisib + ET | NA — Data was not reported for observations including <=5 participants in accordance with hospital data privacy regulations in place at Sinai Health.
  2nd line: ET: number analyzed (Participants) | 21
  2nd line: ET | NA — Data was not reported for observations including <=5 participants in accordance with hospital data privacy regulations in place at Sinai Health.
  2nd line: Chemotherapy: number analyzed (Participants) | 21
  2nd line: Chemotherapy | 6
  3rd line: Palbociclib + ET + goserelin: number analyzed (Participants) | 12
  3rd line: Palbociclib + ET + goserelin | NA — Data was not reported for observations including <=5 participants in accordance with hospital data privacy regulations in place at Sinai Health.
  3rd line: Other CDK 4/6i: number analyzed (Participants) | 12
  3rd line: Other CDK 4/6i | NA — Data was not reported for observations including <=5 participants in accordance with hospital data privacy regulations in place at Sinai Health.
  3rd line: Chemotherapy: number analyzed (Participants) | 12
  3rd line: Chemotherapy | 10

2. Secondary Outcome: Number of Participants Classified According to Type of Treatment Before Introduction of CDK4/6 Inhibitor
Time Frame: From date of ABC/MBC diagnosis until introduction of CDK 4/6 inhibitor(anytime between Jan 2016 to May 2016, approximately 4 months); available data evaluated over approximately 4.5 months of this retrospective study
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study. Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | HR+/HER2- ABC/MBC Participants
Number analyzed (Participants) | 1
Participants | NA — Data was not estimated to protect privacy in accordance with hospital data privacy regulations in place at Sinai Health.

3. Secondary Outcome: Number of Participants Classified According to Type of Treatment After Introduction of CDK4/6 Inhibitor
Time Frame: From date of introduction of CDK4/6 inhibitor until date of death, date of last follow-up or the end of the study period, whichever came first (approximately 33 months); available data evaluated over approximately 4.5 months of this retrospective study
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HR+/HER2- ABC/MBC Participants
Number analyzed (Participants) | 8
Participants | NA — Data was not reported for observations including <=5 participants in accordance with hospital data privacy regulations in place at Sinai Health.

ADVERSE EVENTS:
Time Frame: From date of ABC/MBC diagnosis until date of death, date of last follow-up or the end of the study period, whichever came first (maximum follow-up of 67.6 months); available data evaluated over approximately 4.5 months of this retrospective study.
Arm/Group | HR+/HER2- ABC/MBC Participants
All-Cause Mortality (participants affected / at risk) | 2/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT05770713/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT05770713/SAP_001.pdf